CLINICAL TRIAL: NCT01176994
Title: Safety of Formalin-free Fixatives for In-Vivo Fixation of Skin Lesions.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Michael Kahana, MD, Hillel Yaffe Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HYMC-0016-09
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-07

CONDITIONS: Skin Abnormality
Keywords: Patients with skin lesions that are treated by dermatologists with destructive modalities without histological evaluation.
MeSH Terms: conditions — Skin Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Skin lesions (Experimental): Individuals with skin lesions whose lesions are not sent for histology by dermatologists
  Interventions: Device: Formulations for in-vivo fixation

INTERVENTIONS:
Device: Formulations for in-vivo fixation — Formulations are comprised of non-toxic ingredients used in dermatology.
  Other Names: Formulation ingredients:

SUMMARY:
Existing methods of diagnosing and treating skin lesions are either surgical, which enables an histological diagnosis or destructive (electrodesiccation, liquid nitrogen, laser, caustics) with no possibility of obtaining histology. The ingredients of current formulations for in-vivo skin fixation (Mohs, Solcoderm) are unstable, inconvenient for application and painful - therefore their use was abandoned. The investigators will examine the safety of stable formalin-free formulations for in-vivo fixation of human skin lesions .These formulations were safe and had a rapid onset of fixation effect in in-vivo animal studies.

DETAILED DESCRIPTION:
The formulations are comprised of standard non-toxic laboratory chemicals that are used in various dermatological preparations.

Transition metal salts - Zinc chloride, zinc bromide, zinc iodide,zinc nitrate, zinc sulphate. copper chloride ,copper bromide, copper iodide, copper nitrate, copper sulphate.

Keratolytics - salicylic acid , lactic acid, nitric acid, pyruvic acid,oxalic acid, trichloro acetic acid, phenol, resorcinol,urea .

The solvents and penetration enhancers of the ingredients - Water, ethanol, dimethyl sulfoxide, propylene glycol, glycerol.

Patients with skin lesions that after clinical diagnosis are usually treated by dermatologists with destructive modalities without an histological evaluation will be included in the study. The clinical diagnoses include viral warts, seborrheic warts, skin tags, solar keratoses, fibromata and hemangiomata.

The treated lesions will be located on the trunk and limbs. Lesions on the face will not be included in the study.

The formulations will be infiltrated intra-dermally into the lesions in a maximal volume not exceeding 0.05 ml.

After the achievement of the desired local fixation effect, the lesions will be examined by a pathologist.

The patients will be closely followed-up during the procedure and the degree of possible associated pain will be evaluated. Possible local infection and the degree of scarring will be evaluated until complete healing of the treated area will occur.

The histological result will be informed to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with skin lesions that are not treated with histology

Exclusion Criteria:

* Seriously ill patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Safety | One year
  Infiltration of formulations into skin lesions.
Safety of formulations | One year
  Infiltration of the formulations into skin lesions with resultant in-vivo fixation and the achievement of histological result. Possible local pain, infection and scarring will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel